CLINICAL TRIAL: NCT01365598
Title: Evaluation of the Efficacy and Safety of Primaquine for Clearance of Gametocytes in Uncomplicated Falciparum Malaria in Uganda
Brief Title: Evaluation of the Gametocytocidal Efficacy and Safety of Primaquine in Uncomplicated Falciparum Malaria in Uganda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PQPF912
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Falciparum Malaria
Keywords: malaria; uncomplicated malaria; gametocytocidal drug; gametocytocidal; gametocyte; primaquine; transmission blocking; malaria transmission; sexual parasite; sexual stage; Uganda; Africa
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Primaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Non-active drug
  Interventions: Drug: Primaquine
- Low dose primaquine (PQ1) (Experimental): Lowest experimental dose of primaquine base: 0.1mg/kg
  Interventions: Drug: Primaquine
- Intermediate dose primaquine (PQ2) (Experimental): Intermediate experimental dose of primaquine base: 0.4mg/kg
  Interventions: Drug: Primaquine
- Reference dose primaquine (PQ-R) (Active Comparator): WHO-recommended dose of primaquine base: 0.75mg/kg
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — Single dose of oral primaquine phosphate. Comparator dose is 0.75mg/kg primaquine base. Each experimental arm is a different (reduced) dose of primaquine phosphate. Placebo contains no primaquine phosphate (non-active ingredients only).
  Other Names: primaquine phosphate

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of lower doses of primaquine compared to the dose recommended by the WHO for reducing P. falciparum gametocytes in the infected human host to prevent transmission of falciparum malaria to the anopheles mosquito vector.

DETAILED DESCRIPTION:
A single dose of 0.75mg/kg primaquine base is recommended by the WHO to block transmission of falciparum malaria from infected humans to mosquitoes by clearing gametocytes. However, the optimal dose for safety and efficacy has not been evaluated. Dose-finding data is important because primaquine has a dose-dependent risk of causing haemolysis (destruction of blood cells) in pre-disposed individuals, such as those with G6PD deficiency. G6PD deficiency is most prevalent in malaria-endemic areas. Therefore, it is essential that data on primaquine's safety is available in such areas.

The investigators hypothesise that lower doses of primaquine have a lower risk of adverse effects compared to the WHO-recommended dose, but retain the transmission-blocking efficacy.

The investigators propose to test this hypothesis in a four-arm clinical trial with a non-inferiority design to evaluate the efficacy and a superiority design to evaluate the safety of the WHO dose (0.75mg/kg) and lower doses of primaquine for clearance of P. falciparum gametocytes in children in Uganda. The study will include a pharmacokinetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 1 year and </= 10 years
* Weight over 10kg
* Fever >38 degrees C (tympanic) or history of fever in the last 24 hours
* P. falciparum parasitaemia <500 000/µl
* Normal G6PD enzyme function

Exclusion Criteria:

* Enrolled in another study
* Evidence of severe illness/ danger signs
* Known allergy to study medications
* Haemoglobin < 8g/dL)
* Started menstruation
* Pregnancy or breastfeeding
* Primaquine taken within the last 4 weeks
* Blood transfusion within the last 90 days
* Non-falciparum malaria co-infection

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 468 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mean number of days to gametocyte clearance (gametocyte clearance time, GCT) | 14 days
  Mean number of days per treatment arm for gametocytes to become undetectable using sub-microscopic molecular testing methods (real-time nucleic acid sequence-based amplification, QT-NASBA)and interpolated from measured data points.
Mean (+/- SD) maximal fall in Hb (g/dL) from enrollment to day 28 of follow-up | 28 days
  Mean maximal greatest negative difference in Hb (measured by Hemocue®) from enrollment value per treatment arm over 28 days follow up

SECONDARY OUTCOMES:
Mean (+/- SD) area under the curve of gametocyte density per day during 14 days of follow-up | 14 days
  An estimate of the area under the curve of gametocytes (measured by QT-NASBA) seen over time, averaged per day of follow up (days 0-14) and interpolated from measured data points
Requirement for blood transfusion | 28 days
  Percentage of children receiving blood transfusion per treatment arm during days 0-28
Follow-up day of Hb nadir | 28 days
  Mean day of follow up (day 0-28) per treatment arm of lowest Hb measurement (by Hemocue®)
Incidence of serious adverse events by sign, symptom, laboratory parameter and relationship to taking study drug | 28 days
  Percentage (number) per treatment arm during days 0-28
Incidence of gastrointestinal symptoms after taking study drug | 6 days
  Percentage (number) of children with gastrointestinal symptoms per treatment arm during days 2-7

CONTACTS AND LOCATIONS:
Overall Officials: Alice C Eziefula, MBBS MCRP MRCPath, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Walukuba Health Centre IV, Jinja, Eastern Region, Uganda

REFERENCES:
- [Background] Bousema T, Okell L, Shekalaghe S, Griffin JT, Omar S, Sawa P, Sutherland C, Sauerwein R, Ghani AC, Drakeley C. Revisiting the circulation time of Plasmodium falciparum gametocytes: molecular detection methods to estimate the duration of gametocyte carriage and the effect of gametocytocidal drugs. Malar J. 2010 May 24;9:136. doi: 10.1186/1475-2875-9-136. PMID 20497536
- [Background] Shekalaghe S, Drakeley C, Gosling R, Ndaro A, van Meegeren M, Enevold A, Alifrangis M, Mosha F, Sauerwein R, Bousema T. Primaquine clears submicroscopic Plasmodium falciparum gametocytes that persist after treatment with sulphadoxine-pyrimethamine and artesunate. PLoS One. 2007 Oct 10;2(10):e1023. doi: 10.1371/journal.pone.0001023. PMID 17925871
- [Background] Schneider P, Bousema JT, Gouagna LC, Otieno S, van de Vegte-Bolmer M, Omar SA, Sauerwein RW. Submicroscopic Plasmodium falciparum gametocyte densities frequently result in mosquito infection. Am J Trop Med Hyg. 2007 Mar;76(3):470-4. PMID 17360869
- [Background] Shekalaghe SA, ter Braak R, Daou M, Kavishe R, van den Bijllaardt W, van den Bosch S, Koenderink JB, Luty AJ, Whitty CJ, Drakeley C, Sauerwein RW, Bousema T. In Tanzania, hemolysis after a single dose of primaquine coadministered with an artemisinin is not restricted to glucose-6-phosphate dehydrogenase-deficient (G6PD A-) individuals. Antimicrob Agents Chemother. 2010 May;54(5):1762-8. doi: 10.1128/AAC.01135-09. Epub 2010 Mar 1. PMID 20194698
- [Background] Smithuis F, Kyaw MK, Phe O, Win T, Aung PP, Oo AP, Naing AL, Nyo MY, Myint NZ, Imwong M, Ashley E, Lee SJ, White NJ. Effectiveness of five artemisinin combination regimens with or without primaquine in uncomplicated falciparum malaria: an open-label randomised trial. Lancet Infect Dis. 2010 Oct;10(10):673-81. doi: 10.1016/S1473-3099(10)70187-0. Epub 2010 Sep 9. PMID 20832366
- [Derived] Chang HH, Meibalan E, Zelin J, Daniels R, Eziefula AC, Meyer EC, Tadesse F, Grignard L, Joice RC, Drakeley C, Wirth DF, Volkman SK, Buckee C, Bousema T, Marti M. Persistence of Plasmodium falciparum parasitemia after artemisinin combination therapy: evidence from a randomized trial in Uganda. Sci Rep. 2016 May 20;6:26330. doi: 10.1038/srep26330. PMID 27197604
- [Derived] Eziefula AC, Bousema T, Yeung S, Kamya M, Owaraganise A, Gabagaya G, Bradley J, Grignard L, Lanke KH, Wanzira H, Mpimbaza A, Nsobya S, White NJ, Webb EL, Staedke SG, Drakeley C. Single dose primaquine for clearance of Plasmodium falciparum gametocytes in children with uncomplicated malaria in Uganda: a randomised, controlled, double-blind, dose-ranging trial. Lancet Infect Dis. 2014 Feb;14(2):130-9. doi: 10.1016/S1473-3099(13)70268-8. Epub 2013 Nov 13. PMID 24239324